CLINICAL TRIAL: NCT02230644
Title: RELAX Surgical: Effects of Environmental Design on Pre-surgical Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Music (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SAL1415
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Audio enhanced (Experimental): Enhanced Clinical Environment: participants wait for their operation in the enhanced audio-visual booth.
  Interventions: Other: Enhanced clinical environment
- Other distraction method (Active Comparator): Participants wait for their operation in a booth with another distraction such as the news on television
  Interventions: Other: Other distraction
- Ordinary (No Intervention): Participants wait for their operation in an ordinary, unenhanced booth

INTERVENTIONS:
Other: Enhanced clinical environment — Surgical booths containing artwork and calming background music.
  Arms: Audio enhanced
Other: Other distraction — Such as newspaper, magazine or the news on television
  Arms: Other distraction method

SUMMARY:
Over 4.6 million operations are undertaken each year in England alone. Of these, many patients experience psychological distress, which has negative implications for patient recovery. Indeed, psychological stress, in particular both trait and state anxiety, anger and distress, has been linked with slower wound healing (Broadbent et al., 2003) and more complicated post-operative recovery (Johnston and Wallace, 1990).

However, pre-operative psychological interventions can have significant positive effects on components of of post-operative recovery (Navros et al., 2011; Weinman and Johnston, 1988). In particular, music has been studied in a series of randomised control trials as a way of reducing pre-surgical stress. Studies have shown the effects of music in reducing levels of stress hormones such as cortisol (Leardi et al., 2007) and reducing both heart rate and blood pressure, and have also found music to be more effective than benzodiazepine at reducing pre-surgical anxiety (Bringman et al., 2009).

Chelsea and Westminster Hospital NHS Foundation Trust is a major surgical hospital, performing over 15,000 adult operations annually. Consequently, strategies to reduce patient anxiety and improve experience are amongst the hospital's priorities. A renovation of the Surgical Admissions Lounge is currently underway with plans to incorporate visual arts and music in waiting booths to relax and distract patients. When asked how relaxing they found the space, patients at Chelsea and Westminster Hospital involved in a public consultation rated the current unenhanced waiting area as 5.8/10, but 93% of patients said that relaxing music would help them feel less anxious. This project will test whether music and art in the SAL actively reduce adult patient stress compared to normal unenhanced waiting spaces, with a view to extending the arts interventions to other surgical waiting areas such as the day treatment centre if there are significant positive findings.

DETAILED DESCRIPTION:
Stress can be measured via a number of methods, including both psychological and physiological. This study proposes to examine three signatures of stress in order to triangulate data and achieve a more comprehensive understanding of patients' stress response:

1. Psychological - we will use validated psychological questionnaires including STAI to measure both trait and state anxiety. We will also be using a simple prospective time perception test and a Stroop test to assess whether patients' attention capacity.
2. Physiological - We will use biosensors and bioharnesses to gather electrocardiogram (ECG) data in order to test the complexity loss hypothesis. This hypothesis states that the physiological responses of organisms under constraints (ageing, illness, stress) exhibit grossly reduced dynamics and lose the ability to adopt to the changes in the environment. We will examine whether patients exhibit these reduced dynamics as their operation approaches and whether the arts can be used to increase the complexity of their responses.
3. Biological - we will take two small saliva (spit) samples from patients to test whether levels of stress hormones such as cortisol are elevated in patients, and whether other immune biomarkers such as pro-inflammatory cytokines TNF-alpha and IL-1 are reduced by pre-surgical stress but maintained when music and art are present. Previous research within the field of psychoneuroimmunology suggests that alterations in psychological stress levels have consequences for biological response (Ader, 2007).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Awaiting an operation for which they will have to pass through the surgical admissions lounge.

Exclusion Criteria:

* Wearing of hearing aids (which would prevent participants from wearing the biosensors in their ears)
* Severely impaired sight or hearing (to the level that would affect their ability to participate in the interventions)
* A dementia that would compromise their ability to provide informed consent
* A language barrier that prevents participants from being able to understand the PIS and provide informed consent.
* Pre-surgical sedative administered either prior to or during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Decrease in complexity of physiological response shown from ECG data collected via biosensing electrodes | Over 30 - 90 minutes

SECONDARY OUTCOMES:
Reduction in stress hormones and Th1/Th2 shift in immune biomarkers measured in saliva samples | 30 - 90 minutes

OTHER OUTCOMES:
Reduction in state anxiety measured in psychological scales | 30 - 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Mandic, Principal Investigator — Imperial College London; Aaron Williamon, Study Director — Royal College of Music
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom